CLINICAL TRIAL: NCT05938179
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Study Evaluating the Efficacy and Safety of HS-10353 in Chinese Adults With Depression.
Brief Title: A Study of HS-10353 in Adult Participants With Major Depressive Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10353-201
Record Dates: First submitted 2023-07-03; First posted 2023-07-10 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10353 Capsules (Experimental)
  Interventions: Drug: HS-10353 30mg oral capsules; Drug: HS-10353 50mg oral capsules
- HS-10353 matched-placebo oral capsules (Experimental)
  Interventions: Drug: Placebo for HS-10353 30mg capsules; Drug: Placebo for HS-10353 50mg capsules

INTERVENTIONS:
Drug: HS-10353 30mg oral capsules — HS-10353 30mg oral capsules
  Arms: HS-10353 Capsules
Drug: HS-10353 50mg oral capsules — HS-10353 50mg oral capsules
  Arms: HS-10353 Capsules
Drug: Placebo for HS-10353 30mg capsules — Placebo for HS-10353 30mg capsules
  Arms: HS-10353 matched-placebo oral capsules
Drug: Placebo for HS-10353 50mg capsules — Placebo for HS-10353 50mg capsules
  Arms: HS-10353 matched-placebo oral capsules

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase II clinical study to evaluate the efficacy and safety of continuous oral administration of HS-10353 in Chinese adults with depression.HS-10353 is a new generation of GABAA receptor isomeric modulator developed by our company, which can correct the dysfunction of GABAA receptor function and restore the balance between GABA receptor and NMDA receptor. Oral administration of HS-10353 at night for 14 days is expected to reduce clinical symptoms in patients with depression. As an oral preparation of allopregnenolone analogitics, it has good bioavailability, rapid onset and high safety, and has broad clinical application prospects, which is expected to better meet the treatment needs of clinical depression in China in the future.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years (including the threshold);
* Subjects should have a full understanding of the test content, process and possible adverse reactions, and voluntarily sign an informed consent form (ICF);
* Participants met the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) diagnostic criteria for recurrent depressive disorder (MDD) or single episode MDD without psychotic symptoms, and had an overall HAM-D17 score ≥22;
* No antidepressant therapy has been used during the current episode; Participants who are currently taking antidepressants should be eluted for at least 1 week (or 5 half-lives, whichever is longer) before they can be included in the study.
* Agree to stop using other antidepressants, antianxiety drugs, antipsychotics, mood stabilizers, benzodiazepines sedative and hypnotic drugs during the study treatment;
* According to the investigators, the subjects were generally in good physical condition. During screening, no clinically significant abnormalities were found in physical examination, vital signs, 12-lead electrocardiogram (ECG), laboratory examination (blood routine, blood biochemistry, thyroid function, coagulation function, urine routine, etc.), anterolateral chest X-ray or chest CT.
* Female subjects of reproductive age, serum β-hCG (β-HCG) negative at screening/baseline;
* Subjects must agree to abstain from sex or use other effective contraceptive methods for 30 days from screening until the last dose; Male subjects should agree to refrain from donating sperm from the start of dosing until 6 months after stopping study treatment, and female subjects should agree to refrain from donating eggs from the start of dosing until 6 months after stopping study treatment.

Exclusion Criteria:

* According to the DSM-5 diagnostic criteria, the subject has a current/past history of schizophrenia spectrum or other psychosis, bipolar or related disorders, compulsive and related disorders, trauma and stress-related disorders, dissociation disorders, anorexia or bulimia nervosa, personality disorders, etc.;
* Consistent with the diagnosis of treatment-resistant depression, that is, persistent depressive symptoms after sufficient doses and full courses of two antidepressants are used in a single depressive episode;
* Based on the Columbia-Suicide Severity Assessment Scale (C-SSRS), subjects had a history of suicidal intent/self-harm behavior during the current depressive episode;
* Use of typical/atypical antipsychotics and mood stabilizers during the current depressive episode;
* Previous history of seizures (except convulsions caused by febrile convulsions in children);
* Have a history of severe allergies;
* A history of alcohol or drug dependence/drug abuse (including benzodiazepines, other than nicotine or caffeine) within the last 1 year, or a positive urine drug test at screening;
* Take CYP3A4 suppressant or grapefruit/grapefruit juice, grapefruit/grapefruit, Sevilla orange or products rich in such substances within 14 days prior to screening (or 5 half-lives, whichever is longer);
* Use of CYP inducers such as rifampin, carbamazepine, Ritonavir, enzalutamide, efavirenan, nevirapine, phenytoin, phenobarbital, or St. John's Wort within 14 days (or 5 half-lives, whichever is longer) prior to screening;
* Received modified electroconvulsive therapy (MECT) during the current depressive episode; Or received transcranial magnetic stimulation (TMS), vagus nerve stimulation (VNS), deep brain stimulation (DBS) within 1 week before screening; Or the investigator determines that the subject with the current seizure needs to receive the above treatment;
* Have participated in any clinical trial or taken any clinical trial drug within the last 1 year;
* Women in pregnancy, puerperal period, postpartum 6 months or breastfeeding period, who have planned pregnancy in the near future;
* Poor blood pressure control or abnormal heart rate: at rest, systolic blood pressure (SBP) ≥140 mmHg or < 90 mmHg, diastolic blood pressure (DBP) ≥90 mmHg or < 60 mmHg; Heart rate >100 bpm or <60bpm;
* The presence, in the investigator's judgment, of any surgical condition or condition that is likely to significantly affect drug absorption, distribution, metabolism, or excretion, or that is likely to pose a hazard to participants in the trial; Such as gastrointestinal surgery history (gastrectomy, gastrostomy, enterectomy, etc.), gastroenteritis, gastrointestinal ulcer, gastrointestinal bleeding history; Urinary tract obstruction or dysuria;
* Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis seroreaction (TRUST), human immunodeficiency virus (HIV) antibody test positive;
* Abnormal 12-lead ECG was clinically significant at screening/baseline: QT interval (QTcF) corrected by Fridericia formula had an absolute value of QTcF >450 ms for males and >470 ms for females; If QTcF is prolonged in the first measurement, the average value of 3 consecutive ECGs (10 minutes between each measurement) should be taken to confirm;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN), serum creatinine (Cr) > 1.5 times ULN;
* Patients with diseases that may have clinical significance (such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, skeletal musculoskeletal system, metabolism, endocrine system, skin diseases, blood system diseases, immune diseases and tumors, etc.) are assessed by the researcher as not suitable for participation in this study;
* Any other conditions assessed by the investigator that might interfere with compliance, harm the health of the subject, or interfere with the study outcome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the 17-item HAM-D Total Score at Day 15 | Baseline (BL), Day 15
  The 17-item HAM-D is used to rate the severity of depression in participants who were already diagnosed as depressed. The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 to 2 include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Total HAM-D score can range from 0 to 52, and higher scores indicate severe depression. A negative change from baseline indicates less depression.

SECONDARY OUTCOMES:
Change From Baseline in the 17-item HAM-D Total Score | Baseline, Days 3, 8, 21,28
  The 17-item HAM-D is used to rate the severity of depression in participants who were already diagnosed as depressed. The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 to 2 include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Total HAM-D score can range from 0 to 52, and higher scores indicate severe depression. A negative change from baseline indicates less depression.
Number of Participants Achieving HAM-D Response | Days 3，8，15, 21, and 28
  HAM-D response is defined as a ≥50% reduction in HAM-D score from baseline. The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 to 2 include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Total HAM-D score can range from 0 to 52, and higher scores indicate severe depression.
Number of Participants Achieving HAM-D Remission | Days 3，8，15, 21, and 28
  HAM-D remission is defined as HAM-D total score ≤7. The HAM-D total score comprises a sum of the 17 individual item scores. 8 items scored in a range of 0 to 2 include: Insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following 9 items are scored in a range of 0 to 4: Agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Total HAM-D score can range from 0 to 52, and higher scores indicate severe depression.
Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) | Baseline, Days 15，28
  The 14-item HAM-A is used to rate the severity of symptoms of anxiety. Each of the 14 items is defined by a series of symptoms and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A is calculated by assigning scores of 0 (not present) to 4 (very severe) to each item. Total HAM-A score is calculated as the sum of the 14 individual item scores with a total score range of 0 to 56, where the score of <17 indicates mild severity, 18 to 24 indicates mild to moderate severity, and 25 to 30 indicates moderate to severe severity. A negative change from baseline indicates less severe symptoms.
Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score | Baseline, Days 3, 8, 15，21,28
  The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. Each item is rated on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). Total MADRS score, calculated as the sum of the 10 individual items, ranges from 0 to 60 with a higher score indicating more depression. A negative change from baseline indicates less severe symptoms.
Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score | Baseline, Days 15，28
  The CGI-S uses a 7-point Likert scale to rate the severity of the participant's illness relative to the clinician's past experience with participants who had the same diagnosis. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=extremely ill. A higher score indicates extreme illness/more severity. A negative change from baseline indicates less severe illness.
Number of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE) and Serious TEAE in Treatment and FU Periods | Treatment period: Up to Day 14; FU period: Day 15 to 28
  An adverse event (AE) is any untoward medical occurrence in a participant administered with a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an IP whether or not related to the product. An AE can include any undesirable medical condition, even if no study treatment has been administered. A TEAE is defined as an AE with onset after the start of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study. A serious TEAE is defined as a TEAE that at any dose results in death, is immediately life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or results in a congenital abnormality or birth defect.
Number of Participants With Clinically Significant Abnormalities in Laboratory Measures in Treatment and FU Periods. | Treatment period: Up to Day 14; FU period: Day 15 to 42
  Laboratory parameters include serum chemistry- Alanine aminotransferase: >3x upper limit of normal (ULN); Alanine aminotransferase or aspartate aminotransferase: >3x ULN; Bilirubin: >1.5x ULN, >2x ULN; Calcium: <2.0 millimoles per liter (mmol/L); Gamma Glutamyl Transferase [units per liter (U/L)]: >3xULN; Potassium: >5.4 mmol/L; Sodium: >150 mmol/L; Hematology- Hematocrit : Male <0.385 liter/liter (L/L) and Female <0.345 L/L and Male >0.55 L/L and Female >0.49 L/L; Hemoglobin: Male <115 grams/liter (g/L) and Female <100 g/L; Neutrophils: <1.5 10^9/L.
Number of Participants With Clinically Significant Vital Sign Abnormalities in Treatment and FU Periods | Up to Day 14; FU period: Day 15 to 28
  Vital signs include supine and standing systolic blood pressure (SBP) [millimeters of mercury (mmHg)]: <90, >180, increase and decrease from baseline of >=30; Supine and standing diastolic blood pressure (DBP) (mmHg): Increase and decrease from baseline >=20; Standing heart rate (>120 beats per minute); Orthostatic SBP (>=20); Orthostatic DBP (>=10); Orthostatic hypotension (SBP >=20 and DBP >=10, SBP >=20 or DBP >=10).
Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities in Treatment and FU Periods | Up to Day 14; FU period: Day 15 to 42
  Supine 12-lead ECGs were performed in triplicate and the standard intervals (heart rate, PR, QRS, QT, and corrected QT interval by Fridericia [QTcF]) as well as any rhythm abnormalities were recorded. Criteria for clinically significant ECG abnormalities included QTcF interval (msec)- >500，or longer than 60 msec from baseline
Number of Participants With Suicidal Ideation or Behavior Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) in Double-blind Treatment Period | Up to Day 14; FU period: Day 15 to 42
  Suicidality was monitored during the study using the C-SSRS scale. The C-SSRS includes 'yes' or 'no' responses for 5 questions for assessment of suicidal ideation and behavior. Any suicidal behavior: When response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation: When response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide.
Change From Baseline in SSS Scores in Double-blind Treatment Period | Up to Day 14
  Sleepiness as measured by the Stanford Sleepiness Scale (SSS) has at least two dimensions: activity and sleepiness. The subjects did not perceive the descriptions to be consistent in each dimension. Participants rated their current sleepiness on a scale from 1 to 7. Scores were assigned as follows: feeling energetic, well energetic but not at their best, awake but somewhat loose, having some degree of grogginess, grogginess, sleepiness, wanting to lie down, not trying to stay awake anymore, falling asleep quickly, feeling dreaming.
Change From Baseline in the 20-item Physician Withdrawal Checklist (PWC-20) Total Score | Baseline, Days 15, 21, and 28
  The PWC-20 was used to monitor for the presence of potential withdrawal symptoms following discontinuation of HS-10353. The PWC-20 was made up of a list of 20 symptoms (loss of appetite, nausea-vomiting, diarrhea, anxiety-nervousness, irritability, dysphoric mood-depression, insomnia, fatigue-lethargy-lack of energy, poor coordination, restlessness-agitation, diaphoresis, tremor-tremulousness, dizziness-lightheadedness, headaches, muscle aches or stiffness, weakness, increased acuity [sound, smell, touch, pain], paresthesia, difficulty concentrating and remembering, depersonalization-derealization) that were rated on a scale of 0 (not present) to 3 (severe). The PWC-20 total score was derived as the sum of individual item scores, which ranges from 0 (not present) to 60 (severe). Higher scores indicate more severe withdrawal. A negative change from baseline indicates less severe withdrawal.